CLINICAL TRIAL: NCT03442244
Title: Skin Irritation Trial of LEO 90100 Foam (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Healthy Japanese Subjects
Brief Title: Skin Irritation of LEO 90100 Foam (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: LP0053-1007
Record Dates: First submitted 2018-01-29; First posted 2018-02-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEO 90100 foam (Experimental): Each subject has each of the 2 investigational products applied at the same time on 2 sites on the back. The location on which the treatments are applied is randomised in a double-blinded manner LEO 90100 foam contains Calcipotriol hydrate 52.2 μg/g (equivalent to 50.0 μg/g calcipotriol) plus Betamethasone dipropionate 0.643 mg/g
  Interventions: Drug: LEO 90100 foam
- Vehicle foam (Placebo Comparator): Each subject has each of the 2 investigational products applied at the same time on 2 sites on the back. The location on which the treatments are applied is randomised in a double-blinded manner.
  Foam vehicle does not contain active ingredients
  Interventions: Drug: Vehicle of LEO 90100 foam

INTERVENTIONS:
Drug: LEO 90100 foam — Each subject has each of the 2 treatments applied at the same time on 2 different sites on the back
  Arms: LEO 90100 foam
Drug: Vehicle of LEO 90100 foam — Each subject has each of the 2 treatments applied at the same time on 2 different sites on the back
  Arms: Vehicle foam

SUMMARY:
This trial is looking at whether the LEO 90100 foam causes irritation of the skin in healthy Japanese male adults without psoriasis. A single application of LEO 90100 foam and its vehicle will each be made to 2 body sites in 20 subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent has been obtained.
* Healthy Japanese male subjects.
* Aged 20 to 40 years inclusive.

Key Exclusion Criteria:

* Body Mass Index outside the range 18-25 kg/m²
* Use of any medication (systemic or topical) within 2 weeks of Day 1.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Skin irritation | Up to Day 4
  Skin irritation measured as skin irritation index (summation of clinical scores [ranging from no reaction to blisters] from 49 hrs to 72 hrs after aplication) divided by total number of skin irritation assessments
Photo irritation | Up to Day 4
  Positive ratios calculated from the photo irritation scores

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (1):
- Medical Co. LTA HAKATA clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No